CLINICAL TRIAL: NCT03602079
Title: A Phase I-II, FIH Study of A166 in Locally Advanced/Metastatic Solid Tumors Expressing Human Epidermal Growth Factor Receptor 2 (HER2) or Are HER2 Amplified That Did Not Respond or Stopped Responding to Approved Therapies
Brief Title: Study of A166 in Patients With Relapsed/Refractory Cancers Expressing HER2 Antigen or Having Amplified HER2 Gene
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Klus Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KlusPharma
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Breast Cancer; HER2 Gene Mutation; HER-2 Gene Amplification; HER2 Positive Gastric Cancer; Salivary Gland Cancer; Salivary Gland Tumor; Salivary Gland Carcinoma; Salivary Gland Neoplasms; Lung Cancer; Colo-rectal Cancer; Rare Diseases; Solid Tumor; Recurrent Gastric Cancer; Recurrent Colon Cancer; Recurrent Breast Cancer; Head and Neck Cancer; Head and Neck Carcinoma; Bladder Cancer; Cervical Cancer; Liver Cancer; Bile Duct Cancer; Urologic Cancer; Pancreatic Cancer; Prostate Cancer; Recurrent Prostate Cancer; Rectal Cancer; Recurrent Ovarian Carcinoma; Recurrent Renal Cell Cancer; Rectal Cancer Stage II; Rectal Cancer Stage I; Rectal Cancer Stage III; Skin Cancer; Mouth Cancer; Lip Cancer Stage I; Tongue Cancer; Breast Neoplasm Malignant Primary; Larynx Cancer; Tonsil Cancer; Palate Cancer; Mucoepidermoid Carcinoma; Primary Peritoneal Carcinoma; Mucinous Adenocarcinoma Gastric; Mucinous Breast Cancer Recurrent; Cholangiocarcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Lung Neoplasms; Colonic Neoplasms; Rare Diseases; Stomach Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Liver Neoplasms; Bile Duct Neoplasms; Urologic Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Skin Neoplasms; Mouth Neoplasms; Lip Neoplasms; Tongue Neoplasms; Laryngeal Neoplasms; Tonsillar Neoplasms; Carcinoma, Mucoepidermoid; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I: Dose Escalation (Experimental): Six dose levels have been selected for evaluation in the Phase I part of the study: 0.3, 0.6, 1.2, 2.4, 3.6, and 4.8 mg/kg of A166
  Interventions: Drug: A166
- Phase II: • Cohort 1 (Experimental): HER2 positive (Immunohistochemistry (IHC) 2+ with fluorescence in situ hybridization (FISH) confirmation and Immunohistochemistry (IHC) 3+) breast cancer. Treatment with A166 at recommended Phase II dose.
  Interventions: Drug: A166
- Phase II: • Cohort 2 (Experimental): HER2 positive (Immunohistochemistry (IHC) 2+ with fluorescence in situ hybridization (FISH) confirmation and Immunohistochemistry (IHC) 3+) gastric cancer. Treatment with A166 at recommended Phase II dose.
  Interventions: Drug: A166
- Phase II: • Cohort 3 (Experimental): HER2 low expressing (Immunohistochemistry (IHC) 1+ and IHC 2+ without fluorescence in situ hybridization (FISH) confirmation) breast cancer. Treatment with A166 at recommended Phase II dose.
  Interventions: Drug: A166
- Phase II: • Cohort 4 (Experimental): All cancers other than breast cancer with low HER2 expression (Immunohistochemistry (IHC) 1+ and IHC 2+ without fluorescence in situ hybridization (FISH) confirmation) and HER2 positive (IHC2+ with FISH confirmation and Immunohistochemistry (IHC) 3+) cancers other than breast and gastric cancer. Treatment with A166 at recommended Phase II dose.
  Interventions: Drug: A166

INTERVENTIONS:
Drug: A166 — A166 is an Antibody Drug Conjugate (ADC) targeting HER2 expressing cancer cells.

SUMMARY:
Open-label, Phase I-II, first-in-human (FIH) study for A166 monotherapy in HER2-expressing or amplified patients who progressed on or did not respond to available standard therapies. Patients must have documented HER2 expression or amplification. The patient must have exhausted available standard therapies. Patients will receive study drug as a single IV infusion. Cycles will continue until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
This is an open-label, Phase I-II, first-in-human (FIH) study for A166 as monotherapy in HER2-expressing patients who progressed on or did not respond to available standard therapies. Patients enrolled in this Phase III study must have documented HER2 positivity defined as positive on in situ hybridization (ISH) or next-generation sequencing (NGS) or HER2 expression, defined as at least 1+ by validated immunohistochemistry (IHC) test. The patient must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have ceased to provide clinical benefit for their disease. Patients will receive study drug as a single IV infusion at the prescribed dose level in each treatment cycle. Cycles will continue until disease progression or unacceptable toxicity. The study is divided into 2 parts (Phase I and Phase II).

ELIGIBILITY:
Inclusion Criteria:

Phase I

Patients must meet the following criteria for inclusion into the study:

1. Patients must be able to provide documented voluntary informed consent.
2. Male or female patient ≥ 18 years.
3. Histologically documented, incurable, locally advanced or metastatic cancer.
4. Evaluable or measurable HER2 positive (by ISH or NGS) disease or HER2 expressing disease. HER2 expressing is defined in this protocol as HER2 expression of ≥ 1+ determined by validated IHC.
5. Patients should have no available therapy likely to convey clinical benefit.
6. Granulocyte count ≥ 1,500/μL, platelet count ≥ 100,000/μL, and hemoglobin ≥ 9 g/dL.
7. Serum bilirubin ≤ 1.5 mg/dL, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 × upper limit of normal (ULN), with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) and patients with hepatic and/or bone metastases (alkaline phosphatase ≤ 5 × ULN).
8. Creatinine clearance ≥ 50 mL/min calculated by Cockroft-Gault, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), or Modification of Diet in Renal Disease (MDRD) formulas. Note that 24 hour urine collection is not required but is allowed.
9. ECOG Performance Status ≤ 1.
10. Women of childbearing potential and men must agree to use an approved method of birth control (e.g., hormonal, barrier) while receiving study drug, and for at least 7 months after the last dose of study drug. Women are excluded from birth control if they had had tubal ligation or a hysterectomy.
11. Patients must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and vitiligo.

Exclusion Criteria:

Phase I:

1. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure (New York Heart Association) III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
2. History of Grade ≥ 3 hypersensitivity reaction to trastuzumab.
3. History of any toxicity to trastuzumab that resulted in trastuzumab being permanently discontinued.
4. Symptomatic brain metastases or any radiation or surgery for brain metastases within 3 months of first infusion of study drug.
5. Require supplemental oxygen for daily activities.
6. Documented Grade ≥ 2 peripheral neuropathy.
7. Any chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or biologic therapy treatment within 4 weeks of first infusion of study drug.
8. Any experimental therapy within 4 weeks of first infusion of study drug.
9. Any major surgical procedure within 4 weeks of first infusion of study drug.
10. Diagnosed active liver disease, including viral or other hepatitis, current or history of alcoholism, or cirrhosis. Patients who have positive hepatitis B virus test results due to having been previously vaccinated against hepatitis B, as evidenced by negative hepatitis B surface antigen (HBsAg), negative anti hepatitis B core protein, and positive antibody to the HBsAg (anti-HBs) are not excluded.
11. Have known prior positive test results for human immunodeficiency virus.
12. Uncontrolled hypertension or diabetes.
13. Pregnancy or lactation.
14. Resting corrected QT interval (QTc) > 470 ms at baseline.
15. Left ventricular ejection fraction (LVEF) < 45% determined by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
16. Prior cumulative doxorubicin dose of > 360 mg/m2 or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose | Minimum of 21 days from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Number of patients with dose limiting toxicities

SECONDARY OUTCOMES:
Phase I: Number of patients with Dose Limiting Toxicities | Minimum of 21 days from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Phase I: Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | Every 3 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Phase I: Number of participants who developed measurable anti-drug antibodies | Minimum of 21 days from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Phase I Maximum observed serum or plasma concentration (Cmax). | 84 Days from date of first dose
Phase I Clearance (CL). | 84 Days from date of first dose
Phase I Area under the serum or plasma concentration time curve from 0 to infinity (AUC[0-∞]). | 84 Days from date of first dose
Phase I Terminal phase elimination half life (t½). | 84 Days from date of first dose
Phase I Volume of distribution at terminal phase (Vz). | 84 Days from date of first dose
Phase I Volume of distribution at steady state (Vss). | 84 Days from date of first dose

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon Ahnert, MD, PhD, Study Chair — MD Anderson
Locations (10):
- United States (10):
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Beth Israel Deaconess Medical Center Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Clinical Research Alliance, Inc., Lake Success, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Portland, Oregon
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No